CLINICAL TRIAL: NCT06597253
Title: A Single Centre Study Comparing a Continuous Non-invasive Lactate Sensor Measurement to Standard Invasive Measurements of Venous and Arterial Lactate in Patients Undergoing Elective Coronary Artery Bypass Graft +/- Valve Surgery.
Brief Title: A Single-centre Study Comparing a Non-invasive Lactate Sensor to Standard Invasive Measurements in Patients Undergoing Coronary Artery Bypass Surgery.
Acronym: CONTINUUM L
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 340203
Record Dates: First submitted 2024-08-30; First posted 2024-09-19 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Cardiovascular; Coronary Artery Bypass; Valve Replacement
Keywords: device; coronary artery bypass surgery; lactate; sensor; valve replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lactate Sensor Device Arm (Experimental): Continuous interstitial fluid lactate monitoring using the non-invasive Nemaura Investigational Lactate Device.
  Interventions: Device: Lactate sensor

INTERVENTIONS:
Device: Lactate sensor — Continuous interstitial fluid lactate monitoring using the non-invasive Nemaura Investigational Lactate Device.

SUMMARY:
The main goal of this study is to see how well a non-invasive lactate sensor measures lactate levels compared to standard blood tests. This might reduce the need for frequent blood draws during surgery recovery, and also provide a more comfortable experience for patients. This will also give us information regarding the suitability of the lactate sensor for monitoring other patients - for instance people attending the accident and emergency department with chest pain in which lactate levels may help make a quick diagnosis.

Patients will be approached for this study if they are undergoing routine coronary artery bypass surgery (CABG) or valve replacement surgery. Participants will wear the non-invasive lactate sensor for up to 14 hours, and the readings will be correlated to lactate levels in blood samples. Once the sensor has been removed and the participant has been discharged from their elective surgery admission, the participant has completed the study.

Participation in this study and the data collected from the sensor will help us understand how well it works and how it can be used to improve patient care in the future.

In the future, the data from this new device will be used to train computer algorithms to provide quick responses that could help manage a patients condition, improving future medical care.

DETAILED DESCRIPTION:
Summary of the study design and methodology

The research nurse or doctor will meet with the patient to explain the study and check the following:

Pre-screening: The research nurse, who may also be part of the patients direct care team will look at the records for patients who are attending St Bartholomews hospital for cardiac surgery for grafts and or valve replacement.

Informed Consent: If the patient is eligible and wishes to participate in the study, a qualified individual from the research team will obtain their consent. If the person obtaining the consent is not a doctor, the participant will be given the opportunity to discuss the study with a medically qualified individual.

Screening: The research nurse or doctor will collect demographic information from the patient and ensure the patient meets the study's inclusion and exclusion criteria.

Pre-Surgery Admission: The research nurse will gather details about the patient's medical history and current medications. The patient will have their blood pressure, heart rate, respiratory rate, weight, and height measured, and an ECG performed. Baseline blood samples will be collected as per the standard of care pre-CABG and/ or replacement valve surgery. If the patient agrees to additional blood samples, they will also have samples collected for sex hormone levels.

CABG +/- replacement valve surgery: The patient will then undergo their planned coronary artery bypass graft (CABG) +/- replacement valve surgery as usual.

Sensor Application: After surgery when the patient is settled in Cardiac Intensive Care Unit, the research nurse will place a lactate sensor on the patient's arm. This sensor will continuously measure the patient's lactate levels. The patient may be asleep whilst the sensor is attached.

Blood Sampling: The patient will have hourly blood samples taken through the tubes inserted for their surgery for up to 14 hours to compare with the sensor readings. These samples will include 12 arterial lactate, 12 central venous lactate, and 12 venous troponin samples. Hourly measurements of the patient's blood pressure, heart rate, and respiratory rate will be taken, and any medication changes will be noted. If the patient agrees to additional blood samples, they will also have 6 samples collected for inflammatory profiles and 3 for full blood counts.

Sensor Removal: After 14 hours, the sensor will be removed, and the patient's skin will be checked for any changes, like a rash. The patient will also have their blood pressure, heart rate, and respiratory rate measured, and an ECG performed. Any changes to the patient's medication will be noted.

Follow-Up: The study team will monitor the patient for up to 24 hours after the sensor is removed or until the patient is discharged from the hospital (whichever is earlier). The study team will note any medication changes, measure the patient's blood pressure, heart rate, and respiratory rate, and perform an ECG.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give informed consent
* ≥18 to ≤ 90 years old
* Successful surgery as defined by the below criteria (which will be recorded in the eCRF):

  * Operative Success: The successful completion of coronary artery bypass grafting (CABG) +/- valve insertion with grafts and/or valves
  * Absence of the following complications:
  * Significant bleeding requiring reoperation
  * Evidence of major life-changing stroke

Exclusion Criteria:

* Previous coronary artery bypass grafting
* Recent acute coronary syndrome (within 4 weeks of consent date)
* Heart failure with EF <35% (from TTE or CT from past 6 months - if both available lower value will be used).
* Chronic severe renal failure (estimated eGFR less than 30 mL/min/1.73m2 by the MDRD formula recorded within 6 months of planned consent date)
* Severe anaemia (<10 recorded within 6 months of planned consent date)
* Known or suspected allergies to medical grade silicone adhesives
* Pre-existing skin condition on the upper arm where the device would be applied, including recent burns/ scalds, open wounds or clinically significant skin lesions.
* Patients with implanted medical devices such as pacemakers or other CLMs
* Severe liver cirrhosis (≥ stage III)
* Lymphoedema or pitting oedema at the time of consent
* Pregnancy
* History of ongoing malignant disease
* Hypoalbuminaemia (<35 g/L recorded within 6 months of consent date)
* Those lacking capacity to consent or are deemed vulnerable adults
* Unable to speak English

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-02 (Estimated); Primary Completion 2025-12-12 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Continuous lactate sensor measurement compared venous and arterial blood gas lactate measurements. | 14 hours
  Correlation coefficients describing the strength of association between a non-invasive continuous lactate sensor measurement (using a commercially developed investigational device by Nemaura Pharma Ltd) and local Radiometer ABL 90, venous and arterial blood gas lactate measurements (both absolute and change) measured hourly up to 12 samples within a 14-hour period post-elective CABG +/- valve replacement surgery.
Continuous lactate sensor measurement compared Troponin-T | 14 hours
  Correlation coefficients describing the strength of association between a non-invasive continuous lactate sensor measurement (using a commercially developed investigational device by Nemaura Pharma Ltd) and venous laboratory measurements of high-sensitivity troponin-T measured hourly up to 12 samples within a 14-hour period post-elective CABG +/- valve replacement surgery.

SECONDARY OUTCOMES:
Relationship between arterial and venous lactate measurements | 14 hours
  Correlation coefficients describing the strength of association between arterial and central venous lactate measurements. Up to 12 samples will be taken and compared within a 14-hour period post elective CABG +/- valve replacement surgery.
Evaluate safety of lactate sensor | 24 hours
  Number of patients experiencing adverse reactions or serious adverse reactions to the non-invasive lactate sensor up to 24 hours post application of the device as measured by number of device-related adverse events.
Relationship between arterial and venous lactate and venous troponin measurements | 14 hours
  Correlation coefficients describing the strength of association between arterial/ central venous lactate and venous troponin measurements. Samples taken hourly up to 12 samples within a 14-hour period post-elective CABG +/- valve replacement surgery.

OTHER OUTCOMES:
Exploration of relationship between lactate and inflammatory profiles. | 14 hours
  Determine the time profile and relationship between lactate, markers of inflammation (including hs-CRP, WBC, pro/anti-inflammatory cytokines and chemokines) in venous blood samples.
Exploration of relationship between lactate and sex hormone levels. | 14 hours
  Determine the time profile and relationship between lactate and sex hormones (oestrogen, progesterone, testosterone, FSH, LH, sex hormone binding globulin) in venous blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Anthony Mathur, Study Chair — Queen Mary University of London
Locations (1):
- Barts Health, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided